CLINICAL TRIAL: NCT06106009
Title: A Multi-Part, Phase 1 Study With Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Single- And Multiple-Dose Escalation To Evaluate The Safety, Tolerability, And Pharmacokinetics Of PF-07976016 In Healthy Adult Participants
Brief Title: A Study to Learn How Different Amounts of the Study Medicine Called PF-07976016 Are Tolerated and Act in The Body in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: C5541001
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Intervention Model Description: Part A and B are randomized, double-blinded, sponsor-open, placebo-controlled studies to evaluate safety, tolerability, PK and PD of single and multiple escalating oral doses of PF-07976016 in healthy adult participants, respectively. Part A is a crossover while Part B is a parallel cohort study design. Part A of the study may also evaluate the safety, tolerability and PK in Japanese participants. Part C is an optional open-label, 4-period, fixed-sequence study to evaluate the effect of PF-07976016 on midazolam PK in healthy participants. Part D is an optional sponsor-open, randomized, double-blinded, placebo-controlled multiple dose study of PF-07976016 administered to participants with obesity.
Who Masked: Participant, Investigator
Masking Description: Parts A, B and D are double-blinded and sponsor-open while Part C is open-label.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A Cohort 1 (Experimental): Single dose administration of PF-07976016 and placebo. Participants will receive up to 4 dose levels of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part A Cohort 2 (Experimental): Single dose administration of PF-07976016 and placebo. Participants will receive up to 4 dose levels of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part A Optional Cohort 3 (Experimental): Single dose administration of PF-07976016 and placebo. Participants will receive up to 2 dose levels of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part A Optional Cohort 4 (Experimental): Single dose administration of PF-07976016 and placebo. Participants will receive up to 4 dose levels of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part B Cohort 5 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part B Cohort 6 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part B Cohort 7 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part B Cohort 8 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part B Cohort 9 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part B Optional Cohort 10 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo
- Part C Optional Cohort 11 (Experimental): Single dose midazolam administered alone or in combination with multiple doses of PF-07976016.
  Interventions: Drug: PF-07976016; Drug: Midazolam
- Part C Optional Cohort 12 (Experimental): Single dose midazolam administered alone or in combination with multiple doses of PF-07976016.
  Interventions: Drug: PF-07976016; Drug: Midazolam
- Part D Optional Cohort 13 (Experimental): Multiple dose administration of PF-07976016 or matching placebo.
  Interventions: Drug: PF-07976016; Drug: Placebo

INTERVENTIONS:
Drug: PF-07976016 — Oral solution, oral suspension or solid oral formulation(s)
Drug: Placebo — Oral solution, oral suspension or solid oral formulation(s)
  Arms: Part A Cohort 1; Part A Cohort 2; Part A Optional Cohort 3; Part A Optional Cohort 4; Part B Cohort 5; Part B Cohort 6; Part B Cohort 7; Part B Cohort 8; Part B Cohort 9; Part B Optional Cohort 10; Part D Optional Cohort 13
Drug: Midazolam — Midazolam oral solution
  Arms: Part C Optional Cohort 11; Part C Optional Cohort 12

SUMMARY:
The purpose of this clinical trial is to learn if the study medicine (called PF-07976016) is safe and how it goes in and out of the body in healthy people. The study may also explore if PF-07976016 has the potential to interact with another medicine called midazolam. In addition, the study may explore how PF-07976016 goes into the body of people who have obesity.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female participants of non-childbearing potential aged 18 to 65 years, inclusive, at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. A total body weight >50 kg (110 lb).
3. Parts A, B and C only: BMI of 20-33 kg/m2.
4. Part D only: BMI of 30-40 kg/m2 and may have well controlled hyperlipidemia or hypertension.

Key Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, skin or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Any condition possibly affecting drug absorption.
3. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer). Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.
4. Standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
5. Renal impairment as defined by an estimated glomerular filtration rate of <75 mL/min/1.73 m².
6. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * alanine aminotransferase, aspartate aminotransferase, or bilirubin ≥1.05 × upper limit of normal;
   * fasting plasma glucose > 126 mg/dL;
   * HbA1c ≥6.0% (Parts A,B and C); HbA1c ≥6.5% (Part D);
   * hematuria as defined by ≥1+ heme on urine dipstick;
   * albuminuria as defined by urine albumin/creatinine ratio >30 mg/g.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2024-08-19 (Actual)

PRIMARY OUTCOMES:
Part A: Number of Participants With Treatment Emergent Adverse Events Following Single Doses | Day 1 up to approximately Day 36
Part A: Number of Participants With Clinical Laboratory Abnormalities Following Single Doses | Day 1 up to approximately Day 36
Part A: Number of Participants With Clinically Significant Change in Baseline Vital Signs Following Single Doses | Day 1 up to approximately Day 36
Part A: Number of Participants With Clinically Significant Change from Baseline in Electrocardiogram Findings Following Single Doses | Day 1 up to approximately Day 36
Part B, Parts C and D, if conducted: Number of Participants With Treatment Emergent Adverse Events Following Multiple Doses | Day 1 up to approximately Day 49
Part B, Parts C and D, if conducted: Number of Participants With Clinical Laboratory Abnormalities Following Multiple Doses | Day 1 up to approximately Day 49
Part B, Parts C and D, if conducted: Number of Participants With Clinically Significant Change in Baseline Vital Signs Following Multiple Doses | Day 1 up to approximately Day 49
Part B, Parts C and D, if conducted: Number of Participants With Clinically Significant Change from Baseline in Electrocardiogram Findings Following Multiple Doses | Day 1 up to approximately Day 49

SECONDARY OUTCOMES:
Part A: Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration | Day 1 up to Day 4
Part A: Maximum Observed Plasma Concentration | Day 1 up to Day 4
Part A: Time to Reach Maximum Observed Plasma Concentration | Day 1 up to Day 4
Part A: Area Under the Curve From Time Zero to Extrapolated Infinite Time | Day 1 up to Day 4
Part A: Plasma Half-Life | Day 1 up to Day 4
Part B: Maximum Observed Plasma Concentration | Days 1, 7 and 14
Part B: Time to Reach Maximum Observed Plasma Concentration | Days 1, 7 and 14
Part B: Area Under the Curve From Time Zero to Time Tau | Days 1, 7 and 14
Part B: Plasma Half-Life | Day 14
Part B: Dose Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau | Day 14
Part B: Percent of Dose Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau | Day 14
Part B: Renal Clearance of Drug | Day 14
Part C (if conducted): Maximum Observed Plasma Concentration of Midazolam | Day 1, Day 3 and Day 11
Part C (if conducted): Area Under the Plasma Concentration-Time Curve from Time 0 to the Time of the Last Quantifiable Concentration of Midazolam | Day 1, Day 3 and Day 11
Part C (if conducted): Area Under the Curve From Time Zero to Extrapolated Infinite Time of Midazolam | Day 1, Day 3 and Day 11
Part D (if conducted): Maximum Observed Plasma Concentration of PF-07976016 | Days 1 and 14
Part D (if conducted): Time to Reach Maximum Observed Plasma Concentration of PF-07976016 | Days 1 and 14
Part D (if conducted): Area Under the Curve From Time Zero to Time Tau of PF-07976016 | Days 1 and 14
Part D (if conducted): Plasma Half-Life of PF-07976016 | Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - New Haven, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5541001